CLINICAL TRIAL: NCT05680389
Title: Placebo-controlled, Randomized, Double-blind Study of Minocycline for Sporadic and Hereditary Cerebral Amyloid Angiopathy
Brief Title: Antibiotics Against Amyloid Angiopathy
Acronym: BATMAN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Marieke JH Wermer, MD, Prof Wermer, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P19.110; 2019-004786-41 (EudraCT Number)
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline (Experimental): 100 mg twice daily for 3 months
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): twice daily for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — 100 mg twice daily for 3 months
  Arms: Minocycline
Drug: Placebo — twice daily for 3 months
  Arms: Placebo

SUMMARY:
We will perform a randomized clinical trial with minocycline. Minocycline is an antibiotic of the tetracycline family and known to modulate inflammation, gelatinase activity and angiogenesis, which we know are central mechanisms in CAA-pathology. Our aim is to prove in a randomized clinical trial in a translational setting that minocycline treatment (duration 3 months) can decrease markers of neuroinflammation and the gelatinase pathway in the cerebrospinal fluid (CSF) of persons with D-CAA (n=30) and sporadic-CAA (n=30).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years for D-CAA and age ≥55 years for sporadic-CAA
* Probable-CAA according to the Modified-Boston-Criteria or genetically proven D-CAA
* ≤ 2 ICH (occurrence of ICHs at least 1 year ago) and presence of ≥ 2 lobar microbleeds +/-cortical superficial siderosis
* Written informed consent

Exclusion Criteria:

* Previous allergic reactions to minocycline
* Modified Rankin Score ≥3
* Contraindications, such as:
* Contraindications for 7T MRI as determined by the 7Tesla safety committee. Examples of possible contra-indications are: claustrophobia, pacemakers and defibrillators, nerve stimulators, intracranial clips, intraorbital or intraocular metallic fragments, cochlear implants, ferromagnetic implants, hydrocephalus pump, intra-uterine device, permanent make-up, tattoos above the shoulders. In case of specific contra-indications for 7T a 3T will be made instead. - Specific contraindications for checkerboard fMRI: seizure within prior year, photosensitive epilepsy, noncorrectable visual impairment. - Contraindications for lumbar puncture: compression of the spinal cord, signs and symptoms of increased intracranial pressure, local infections of the skin at the puncture site, a coagulopathy or thrombocytopenia (<100). (Use of acetylsalicylic acid, NSAIDs, COX2 inhibitors or low-molecular-weight heparin are no contraindications for lumbar puncture.)
* Pregnancy/breast feeding
* Liver/renal failure
* Use of antibiotics <1 month
* SLE or other diseases known to generate inflammatory responses
* Previous/current/planned use of retinoids (since this is related to increasing risk of increased intracranial pressure)
* Current use of anaesthetics like methoxyflurane, agents inhibiting peristalsis, barbiturates, carbamazepine or fenytoïne

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
inflammatory, vessel integrity and gelatinase pathway associated biomarkers in CSF | 3 months
  IL6, MCP-1, IBA-1, MMP2/9, and VEGF

SECONDARY OUTCOMES:
safety and tolerability of minocycline | 3 months
  side effects and adverse events
progression of hemorrhagic markers on 7T MRI before and after treatment | 3 months
  cSS, cortical microbleeds

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voigt S, Koemans EA, Rasing I, van Etten ES, Terwindt GM, Baas F, Kaushik K, van Es ACGM, van Buchem MA, van Osch MJP, van Walderveen MAA, Klijn CJM, Verbeek MM, van der Weerd L, Wermer MJH. Minocycline for sporadic and hereditary cerebral amyloid angiopathy (BATMAN): study protocol for a placebo-controlled randomized double-blind trial. Trials. 2023 Jun 5;24(1):378. doi: 10.1186/s13063-023-07371-4. PMID 37277877